CLINICAL TRIAL: NCT01986543
Title: Interaction Between High Dose Rifampicine and Efavirenz in Pulmonary Tuberculosis and HIV Co-infection
Acronym: RIFAVIRENZ
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12292 RIFAVIRENZ
Record Dates: First submitted 2013-11-12; First posted 2013-11-18 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Tuberculosis; HIV
Keywords: Pharmacokinetic
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): 8 weeks R20mg/Kg + HZE and efavirenz 600mg
  Interventions: Drug: drug administration
- Arm 2 (Experimental): 8 weeks R20mg/Kg + HZE and efavirenz 800mg
  Interventions: Drug: drug administration
- Standard arm (Active Comparator): 8 weeks R10mg/Kg + HZE and efavirenz 600mg
  Interventions: Drug: drug administration

INTERVENTIONS:
Drug: drug administration

SUMMARY:
We propose a first interaction study between efavirenz (EFV) and R20mg/Kg taking into consideration the absence of data about R induction at this dose. Due to an important inter-patient variability of the CYP2B6 polymorphism, the EFV pharmacokinetic (Pk) will be compared in same patients with and without TB treatment.

The main objective is to compare the Pk parameters of EFV in HIV-TB co-infected patients, with and without TB treatment, using R at 10 and 20mg/Kg/day and EFV at 600 and 800mg/day.

DETAILED DESCRIPTION:
Justification: In vitro and animal studies have shown that increasing the dose of rifampicin (R) improves the R sterilising effect. If a similar effect can be demonstrated in the clinical setting, this could allow shortening treatment duration from 6 to 4 months, with good tolerance. Several phase 2 trials in HIV-negative patients are ongoing. We propose a first interaction study between efavirenz (EFV) and R20mg/Kg taking into consideration the absence of data about R induction at this dose. Due to an important inter-patient variability of the CYP2B6 polymorphism, the EFV pharmacokinetic (Pk) will be compared in same patients with and without TB treatment.

Principal objective: To compare the Pk parameters of EFV in HIV-TB co-infected patients, with and without TB treatment, using R at 10 and 20mg/Kg/day and EFV at 600 and 800mg/day.

Secondary objectives: To describe the Pk parameters of R and isoniazid (H); the TB treatment réponse (Mycobacterium tuberculosis culture conversion after 8 weeks(w) and cure after 24w) ; the virological response; the occurrence of severe adverse events, especially hepatic and neurological events; the treatment adherence; the genes involved in the EFV metabolism of EFV, R and H, and its relation with the Pk parameters.

Primary endpoint: AUC0-24, Cmax, Cmin, Tmax of EFV after 4w of TB treatment + ARV, and 4w after interruption of TB treatment.

Study design : phase 2 randomized, open label 3 arms therapeutic trial:

* Arm 1 : 8 weeks R20mg/Kg + H + pyrazinamide(Z)+ ethambutol(E) and EFV600mg/J + tenofovir-lamivudine
* Arm 2: 8 weeks R20mg/Kg + H+Z+E and EFV800mg/J + tenofovir-lamivudine
* Standard arm : 8 weeks R10mg/Kg + H+Z+E and EFV600mg/J + tenofovir-lamivudine

The ARV treatment will be initiated 4 weeks after starting TB treatment. After 8 weeks, all patients will receive 16 weeks of H+R with R at 10mg/Kg/day and EFV at 600mg/day. Treatment will be observed at home by a domiciliary treatment monitor (DTM). Patients will be followed during 28 weeks after starting TB treatment: weekly visit during first 8 weeks and then every 4 weeks.

Pk sampling for EFV, R and H will be at w2 (Pk1), w8 (Pk2) and w28 (Pk3). Liver function test and full blood count will be measured after 2, 4 and 8 weeks; sputum culture for TB at baseline and w8; HIV-1 RNA at baseline, w4, w12 and w24 and CD4 count at baseline and w24.

Eligibility criteria: > 18 years old; previously untreated pulmonary TB; Xpert confirming Mtb susceptible to R; body weight >45Kg; CD4 between 50 and 250cells/mm3; Karnofsky score >80%; ALAT/biluribin <5xULN; no grade 4 clinical/biological sign; no pregnancy + barrier contraception; agree to participate and sign a consent form.

Randomisation block, 1:1:1. Sample size: 28 patients to show that the reduction of AUC of EFV with R20mg/Kg vs no R is not greater to 30%, with 20% expected reduction. Same number per study arm and 20% increase for patients' withdrawals or lost to follow-up resulting in a total of 105 patients.

Site: Mbarara (Uganda)

ELIGIBILITY:
Inclusion Criteria:

* Aged of 18 years or more
* Diagnosis of new pulmonary tuberculosis confirmed by a XpertMTB/RIF test
* Positive HIV antibody test, naïve of ART with CD4 cell count between 50 and 250cells/mm3
* For women of childbearing age, to have a negative urine test for pregnancy on the day of enrolment and to accept to take a barrier contraception during the period of the trial
* Participants well enough to receive ambulatory treatment
* Weight > 45Kg
* Home address readily accessible
* Participants providing informed consent to participate in the trial

Exclusion Criteria:

* Rifampicin drug resistance based on the XpertMTB/RIF result confirmed by the GenotypeMTBDRplus assay
* Concomitant opportunistic infection requiring additional infectious medication
* Karnofsky score <80%
* ALAT or bilirubin > 5.0 x ULN (hepatitis grade 3 or 4)
* Haemoglobin < 7.5g/dL (grade 3 or 4)
* Grade 4 clinical sign or biological result according to the ANRS for grading the intensity of adverse events
* Patient not able to give his informed consent or is unlikely or unable to cooperate with sampling procedures
* Patient suffering of psychiatric illness, which may prevent follow-up according to the protocol
* Patients receiving or requiring medications that may interfere with study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Efavirenz through concentration before drug intake (Cmin); maximal concentration (Cmax); time to achieve the Cmax (Tmax) and area under the curve of concentrations vs time at steady state during a 24-hour dosing interval (AUC0-24) | Week 8
Efavirenz Cmin; Cmax; Tmax; AUC0-24 | Week 28

SECONDARY OUTCOMES:
Pharmacokinetic parameters of R and H (Cmin, Cmax and AUC0-24) | Week 2
Pharmacokinetic parameters of R and H (Cmin, Cmax and AUC0-24) | Week 8
Mycobacterium tuberculosis culture of sputum | week 8
Plasma HIV-1 RNA | week 28
Grade 3 and 4 adverse events | 0-28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: BONNET Maryline, MD, Principal Investigator — Epicentre MSF
Locations (1):
- Mbarara Research Base, Mbarara PO Box 1956, Mbarara, Uganda